CLINICAL TRIAL: NCT07319351
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate Safety and Preliminary Efficacy of TISA-818-Inj in Patients With Acute Respiratory Distress Syndrome
Brief Title: Safety and Preliminary Efficacy of TISA-818 Injection in Patients With Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EnliTISA (Shanghai) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TISA-818-23201
Record Dates: First submitted 2025-12-07; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 6 mg b.i.d TISA-818-Inj (Experimental)
  Interventions: Drug: TISA-818-Inj
- 12 mg q.d. TISA-818-Inj (Experimental)
  Interventions: Drug: TISA-818-Inj
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TISA-818-Inj — 6 mg b.i.d TISA-818-Inj
  Arms: 6 mg b.i.d TISA-818-Inj
Drug: TISA-818-Inj — 12 mg q.d. TISA-818-Inj
  Arms: 12 mg q.d. TISA-818-Inj
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase II clinical study of TISA-818-Inj in patients with ARDS to evaluate the safety, preliminary efficacy, and population PK (Pop PK) profile of TISA-818-Inj in adult ARDS patients.

Totally 60 subjects with ARDS are planned to be included in this study. Subjects will be assigned to the 6 mg twice daily (BID) TISA-818-Inj group, 12 mg once daily (QD) TISA-818-Inj group, or the placebo control group in a 1:1:1 ratio using a stratified block randomization method.

This study includes a screening period (Day -3 to Day -1), a treatment period (Day 1 to Day 14),a short-term follow-up period (Day 15 to Day 60) and a long-term follow-up period (Day 61 to Day 180). Consenting subjects will be screened for eligibility, according to study-specific inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion criteria

1. Voluntarily participate in the clinical study, and patients themselves or their guardians fully understand and are informed of the study and sign the informed consent form, agree to follow and be able to complete all study procedures;
2. Male or female subject age 18-80 years of signing the informed consente;
3. Meets all the following diagnostic criteria:

   1. Timing: Within 1 week of a known clinical insult or new or worsening respiratory symptoms;
   2. Chest imaging: Chest radiography or CT scan showing bilateral opacities - not fully explained by effusions, lobar/lung collapse, or nodules;
   3. Origin of edema: Respiratory failure not fully explained by cardiac failure or fluid overload. Need objective assessment to exclude hydrostatic edema if no risk factor present;
   4. Oxygenation: PaO2/FiO2 ≤ 300 mmHg with PEEP ≥ 5 cm H2O or PaO2/FiO2 ≤ 300 mmHg with high flow nasal oxygen ≥30 L/min;
4. ARDS caused by pneumonia infection;
5. C-reactive protein (CRP) level is higher than the upper limit of normal (ULN) value;
6. Be able to receive the investigational drug within 72 hours after the first diagnosis of the ARDS;
7. Men and women of childbearing potential (women of childbearing potential include premenopausal women and those within 2 years of menopause) who are willing to use highly effective contraception (condom, contraceptive sponge, gel, film, intrauterine device, oral or injected contraceptives, subcutaneous implants, etc.) from signing the informed consent form through 6 months after the last dose of the investigational drug.

Exclusion criteria

1. ARDS caused by drowning or COVID-19;
2. Be allergic to the test drug or excipients;
3. Have an expected survival of ≤ 72 hours as judged by the investigator;
4. Have other current or previous serious pulmonary disease at screening, including but not limited to WHO Class III or IV pulmonary hypertension, chronic lung disease requiring long-term oxygen therapy, or previous lung transplantation;
5. Have a current or previous active cardiovascular disease at screening, including but not limited to Chronic heart disease (New York Heart Association functional class IV), episodes of cardiac arrest or acute myocardial infarction within 4 weeks before screening;
6. Severe hemodynamic instability at screening (defined as norepinephrine dose > 0.5 μg/kg/min or dopamine dose > 20 μg/kg/min);
7. Chronic hemodialysis and known severe renal impairment (creatinine clearance rate<30 mL/min, appendix 8);
8. The following laboratory abnormal values exist:

   * Bone marrow function: platelet count <30 × 109/L, hemoglobin<7.0 g/dL;
   * Liver function: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times the ULN value and serum bilirubin (T-Bil) >2 times the ULN,;
9. Receiving extracorporeal membrane oxygenation (ECMO), continuous renal replacement therapy (CRRT), plasma exchange, hemoperfusion/adsorption, or any other forms of extracorporeal life support at randomization;
10. Have scheduled or anticipated surgery within 28 days after the first administration;
11. Pregnant or lactating women;
12. Those who have used ulinastatin, thymalfasin, Xuebijing, sivelestat sodium and montelukast sodium within 24 hours before starting treatment or systemic treatment with immunosuppressants or other anti-inflammatory agents within 14 days prior to the first administration;
13. The dosage of methylprednisolone used before treatment is > 40 mg/day (or equivalent glucocorticoid) for more than 7 days or the dosage of methylprednisolone used is > 280 mg within 7 days before starting treatment;
14. Those who use any other investigational medicinal product within 28 days before starting treatment;
15. The presence of active pulmonary tuberculosis determined by the investigator, or other active infections that investigator believes may affect the participation or affect the outcome;
16. Patients with malignant tumors requiring treatment in the past 2 years or during screening (skin basal-cell carcinoma, breast/cervical carcinoma in situ, papillary thyroid carcinoma, and other malignant tumors that have been treated and have been effectively controlled in the past 2 years or at the time of screening, can be included in this study if they are judged suitable by investigator);
17. Judgement by the investigator that participation in this study is not in line with the patient's best interests or other conditions that make participation in this study inappropriate, such as poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events as coded by MedDRA and assessed by CTCAE v5.0 | Up to 60 days
  Number of participants with TEAEs following administration of TISA-818 injection

SECONDARY OUTCOMES:
Ventilator-free days (VFD) | Up to 28 days
  The number of days within 28 days that do not require invasive mechanical ventilation, non-invasive mechanical ventilation, or high-flow oxygen therapy.
Days without non-invasive mechanical ventilation/ high-flow oxygen therapy | Up to 28 days
  Number of days for patients need non-invasive mechanical ventilation/ high-flow oxygen therapy.
Days without invasive mechanical ventilation | Up to 28 days
  Number of days without invasive mechanical ventilation.
oxygenation index (PFR) | Day 3, 7, 10, 14, 21, 28
  Changes in PFR compared to baseline and PFR improvement rate.
Plasma population pharmacokinetic (Pop PK) characteristics of TISA-818-Inj in patients with ARDS | Up to 28 days
  For PK analysis, blood samples will be collected before and up to 12h after administration at day 1 and day 5. Blood samples will be collected 30min before administration at day 3, 4, 6, 7, 10 and 14. Blood samples will be collected at day21 and day 28.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The results of this trial will not be published in the International Committee of Medical Journal.